CLINICAL TRIAL: NCT01726426
Title: Modulation of Anaerobic Gut Bacteria in Palmer Arsenical Keratosis Patients by Supplementation With Probiotics
Brief Title: Modulation of Anaerobic Gut Bacteria of Arsenicosis Patients by Probiotics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Prof. Mir Misbahuddin, Prof. and Chairman, Department of Pharmacology, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BSMMU-001-CT
Record Dates: First submitted 2012-11-03; First posted 2012-11-15 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-05

CONDITIONS: Chronic Arsenic Poisoning
Keywords: Chronic arsenic poisoning; Palmer arsenical keratosis
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Patients of palmer arsenical keratosis (Experimental): Probiotics Capsule (Lactobacillus- 2 billion, Bifidobacterium- 1 billion, fructo-oligosaccharide): 1 capsule twice daily orally for 12 weeks
  Interventions: Dietary Supplement: Probiotic
- Arsenic exposed controls (Active Comparator): Probiotics Capsule (Lactobacillus- 2 billion, Bifidobacterium- 1 billion, fructo-oligosaccharide): 1 capsule twice daily orally for 12 weeks
  Interventions: Dietary Supplement: Probiotic
- Heathy volunteers (Active Comparator): Probiotics Capsule (Lactobacillus- 2 billion, Bifidobacterium- 1 billion, fructo-oligosaccharide): 1 capsule twice daily orally for 12 weeks
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Probiotic — Each capsule Probiotics (Lactobacillus- 2 billion, Bifidobacterium- 1 billion, fructo-oligosaccharide): 1 capsule twice daily orally for 12 weeks

SUMMARY:
The role of anaerobic bacteria in the pathogenesis of palmer arsenical keratosis is not known. This can be evaluated by administering probiotics. Thirty patients from an arsenic affected area will be provided two probiotics capsules per day orally for 12 weeks and stool samples will be collected for qualitative and quantitative analysis of anaerobic bacteria. Similar number of arsenic exposed controls and healthy volunteers from the same area will be included with similar protocol for comparison. Like aerobic bacteria, anaerobic bacteria may be modulated by probiotics in arsenicosis patients.

DETAILED DESCRIPTION:
Recent study done by our laboratory shows that there are reduction in the number of E. coli in the gut of patients with arsenical keratosis which is increase by the administration of probiotics (manuscript is preparing). However, E.coli contribute only about 0.1% of the total gut bacteria. It is not known whether anaerobic bacteria play an important role in the pathogenesis of arsenical keratosis. This can be evaluated by administering probiotics. Thirty patients of moderate arsenical palmer keratosis from an arsenic affected area will be recruited on the basis of inclusion and exclusion criteria. They will be provided two probiotics capsules per day orally for 12 weeks. Water sample will be collected before starting the study for confirming the diagnosis. Stool samples will be collected twice (before and after completion of the study) for qualitative and quantitative analysis of anaerobic bacteria. Similar number of arsenic exposed controls (30) and healthy volunteers (30) from the same area will be included in this study and they will be provided probiotics capsules with similar dosage and duration. Like aerobic bacteria, anaerobic bacteria may be modulated by probiotics in arsenicosis patients.

ELIGIBILITY:
Inclusion Criteria (Patients):

* history of taking arsenic contaminated water (>50 ppb) for more than 6 months
* patients having moderate arsenical keratosis present on palm of the hand
* patients those voluntarily agree to participate

Inclusion Criteria (Arsenic exposed controls):

* family member of the patient
* drinking arsenic contaminated water from the same source as patient
* those voluntarily agreed to participate
* no sign/symptoms of palmer keratosis

Inclusion Criteria (Healthy volunteers):

* drinking arsenic safe water <50 ppb)
* those voluntarily agreed to participate

Exclusion Criteria:

* pregnancy
* lactating mother
* patient receiving treatment of arsenicosis
* any other chronic disease like tuberculosis, diabetes, asthma

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2013-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number of pathogenic anaerobic bacteria in stool | 0 weeks (baseline), 12 weeks (end)
  Number of pathogenic anaerobic bacteria in the stool of patients will be decrease in comparison to arsenic exposed controls and volunteers after 12 weeks supplementation with probiotics.

SECONDARY OUTCOMES:
Arsenic level in stool | 0 week (baseline), 12 weeks (end)
  Arsenic level in the stool of patients will be increased in comparison to arsenic exposed controls and healthy volunteers. Arsenic level will be estimated using Atomic Fluorescence spectrometer.
Changes in palmer keratosis following supplementation | 0 week (baseline), 12 weeks (end)
  There will be improvement of moderate palmer keratosis following supplementation with probiotics.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pharmacology, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh